CLINICAL TRIAL: NCT06064370
Title: Side-specific Factors for Intraoperative Hemodynamic Instability in Adrenalectomy for Pheochromocytoma. A Comparative Analysis
Brief Title: Side-specific Factors for Intraoperative Hemodynamic Instability in Pheochromocytoma
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: adrenalectomy
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: adrenalDisease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic right adrenalectomy: laparoscopic right adrenalectomy for pheochromocytoma
  Interventions: Procedure: laparoscopic adrenalectomy
- laparoscopic left adrenalectomy: laparoscopic left adrenalectomy for pheochromocytoma
  Interventions: Procedure: laparoscopic adrenalectomy

INTERVENTIONS:
Procedure: laparoscopic adrenalectomy — laparoscopic adrenalectomy for pheochromocytoma

SUMMARY:
The performance of adrenalectomy for pheochromocytoma (PHEO) presents significant challenges due to the presence of elevated intraoperative hemodynamic instability (HI) and conversion risk. The objective of this study was to conduct a comparative analysis of the occurrence and determinants of perioperative hypotension (HI) and conversion in left-sided (LLA) and right-sided (RLA) transabdominal laparoscopic adrenalectomy (TLA).

DETAILED DESCRIPTION:
Pheochromocytoma (PHEO) is a malignancy characterized by the production of catecholamines from chromaffin cells located in the adrenomedullary system. The prevalence of PHEO in the general population ranges from 0.05% to 0.1%, however it is more prevalent among those with hypertension. The clinical presentation exhibits a spectrum that spans from asymptomatic to abrupt mortality. Minimally invasive laparoscopic adrenalectomy (LA) has emerged as a prominent technique in adrenal illness surgery due to its reduced surgical morbidity and death rates, making it the favored method in this field. The initial exploration of transperitoneal laparoscopic adrenalectomy (TLA) was conducted by Gagner et al. The LA procedure encompasses many transabdominal and retroperitoneal techniques, whereas TLA is favored by surgeons due to its well-known anatomy and expansive working area. Nevertheless, PHEO surgery remains a formidable task for surgeons and anesthesiologists due to its established correlation with hemodynamic instability (HI), resulting in symptoms such as abrupt hypertension or tachycardia, as well as severe and protracted hypotension following tumor excision. Skilled surgeons and anesthesiologists enhance the outcomes and reduce the occurrence of hypotension. The research has documented a multitude of additional risk factors associated with HI. The observed variability could perhaps be attributed to the lack of consistent anesthesiological and surgical protocols, as well as variations in the definitions of HI. Laparoscopic adrenalectomy does not have any absolute contraindications. However, it is worth noting that up to 20% of patients may need to undergo conversion to an open procedure. There has been no specific evaluation of the incidence and risk factors of perioperative hypotension (both intraoperative and postoperative) and conversion rate in a large group of patients undergoing laparoscopic right adrenalectomy (LRA) or laparoscopic left adrenalectomy (LLA) for managing pheochromocytoma resection.

ELIGIBILITY:
Inclusion Criteria:

- patients >18 years, both sex with unilateral PHEO of any size who underwent TLA

Exclusion Criteria:

* Patients who have undergone initial open adrenalectomy, various surgical procedures during total laparoscopic adrenalectomy (TLA), complete adrenalectomy,

bilateral PHEOS bleeding diathesis, skeletal deformity, pregnancy, previous homolateral abdominal surgery, missing data, questionable preoperative diagnosis, inherited PHEO, or recurrent PHEO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 271 patients (n = 271) were involved in the study and subsequently separated into two groups: LRA (n = 122) and LLA (n = 149).
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
hemodynamic instability | intraoperative and immediate postoperative
  incidence of hemodynamic instability

SECONDARY OUTCOMES:
conversion rate | intraoperative
  incidence of conversion

IPD SHARING:
Plan to Share IPD: No